CLINICAL TRIAL: NCT00015288
Title: PK0496 Pharmacokinetics of Buprenorphine
Brief Title: Buprenorphine and Naloxone Combination Study - 10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: New York MDRU (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-5-0013-10; Y01-5-0013-10
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1998-08

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
The purpose of this study is to examine pharmacokinetics and dose proportionality of sublingual tablets containing varying doses of buprenorphine and naloxone.

DETAILED DESCRIPTION:
The objective of this study is to examine pharmacokinetics and dose proportionality of sublingual tablets containing varying doses of buprenorphine and naloxone.

ELIGIBILITY:
Inclusion Criteria:

Male/Female between the ages of 21 and 45. Within 15% of ideal body weight. No oral pathology that would interfere with the sublingual absorption of the medication. Experienced in the use of opiates but not dependent.

Exclusion Criteria:

LFT's exceeding than 3x's normal. History of seizure. Opiate dependent.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-11

PRIMARY OUTCOMES:
Physiological measures
Measurements of buprenorphine and naloxone in plasma
Subjective symptoms measures

CONTACTS AND LOCATIONS:
Overall Officials: John Rotrosen, M.D., Principal Investigator — New York MDRU
Locations (1):
- New York MDRU, New York, New York, United States